CLINICAL TRIAL: NCT03489655
Title: Helping Chicago's Westside Adults Breathe and Thrive: Long Term Effectiveness of a Healthy Homes Approach to Improving Respiratory Health
Brief Title: Helping Chicago's Westside Adults Breathe and Thrive
Acronym: HCWABT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sinai Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ILHHU0029-15; ILHHU0029-15 (Other Grant/Funding Number: U.S. Department of Housing and Urban Development)
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Asthma
Keywords: Healthy Homes; Asthma; Community Health Worker
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maintenance Phase Intervention (Experimental): Participants receive a phone-based Community Health Worker (CHW) intervention in addition to bi-monthly data collection calls with a research assistant.
  Interventions: Behavioral: Maintenance Phase Intervention
- Maintenance Phase Control (No Intervention): Participants receive no further interventions, but have bi-monthly data collection calls with a research assistant.

INTERVENTIONS:
Behavioral: Maintenance Phase Intervention — The CHW will utilize motivational interviewing techniques over phone calls to reinforce all asthma education provided in the AI phase, including asthma basics, triggers and reduction strategies, purpose of medications, and steps for proper medication use. The CHW will identify barriers the participant is facing in management of their asthma and set goals to overcome them. The CHW will encourage regular visits with the Primary Care Physician and assist with referrals for other medical and social services, as needed. CHWs will check-in with participants via phone, monthly for the first 6 months and bi-monthly in the remaining 6 months Participants will receive bi-monthly data collection follow-up phone calls by a Research Assistant.
  Arms: Maintenance Phase Intervention

SUMMARY:
Adults with asthma living in Chicago's West and Southwest side who completed the home-based Community Health Worker (CHW) intervention called Helping Chicago's Westside Adults Breathe and Thrive (HCWABT I) after October 2015 were eligible to participate in a randomized control trial called HCWABT II, which will evaluate the long-term impact of the intervention on their asthma control, asthma severity, healthcare use, and asthma-related quality of life. Participants are randomly assigned to an intervention arm, where they continue to receive occasional (monthly or bimonthly) contact from the CHW who served them during HCWABT I. or a control arm, where they no longer receive contact from the CHW. Members of both groups receive monthly data collection calls from a Research Assistant. We hypothesize that participants in the control arm will experience sustained improvements in asthma outcomes as compared to their pre-HCWABT I levels and that participants in the CHW intervention arm will continue to improve in asthma control severity, quality of life, and healthcare use.

DETAILED DESCRIPTION:
Participants who enroll into HCWABT II will be randomized into one of two study arms: MPI or MPC. In order to randomly choose which arm participants will be enrolled into, the RA will select an envelope prior to the 12-Month visit that will tell them which arm to consent the participant into. A total of 68 envelopes will read MPI and 68 envelopes will read MPC. If a participant declines the maintenance phase, that envelope will be recycled for a future drawing.

All data will be stored in a password-protected database on Sinai's secure server. Data will be de-identified, except for one data collection tool, the Personal Data Sheet, which will contain the participant's personal information along with their study ID. This information will be kept in a separate password protected database. All data will be archived. Paper files will be saved for a minimum of seven years in a secure locked facility. Electronic data will be saved indefinitely, but will always remain password protected and stored on a secure server hosted by Sinai's Information Systems Department. De-identified data will be available to researchers who wish to use it through a data agreement approved by both institutions. Findings will be widely disseminated. The dissemination plan is discussed in Rating Factor 5.

Baseline characteristics will be compared between participants who complete the entire intervention and follow-up period, and those who are either lost to follow-up or dropout, to assess the effect of selection bias. Dropout and completion rates will be reported. Screening-to-enrollment ratios will be calculated from screening data. Frequencies, means and medians, as appropriate, will be calculated for each outcome variable at baseline and over the follow-up period associated with that outcome. The effect of the 12-month AI will be evaluated using pre-posttest methods with each participant serving as his/her own historical control. Participants enrolled in Maintenance RCT will be both evaluated against their own historical data as well as the data of the other arm of the study. A cost effectiveness analysis will also be conducted using process measures, including staff time, materials, referrals and time spent on various intervention activities in order to calculate program-specific costs. Non-parametric tests will be used to assess whether changes between baseline and follow-up are statistically significant. In cases where the degree of difference is important, such as when comparing differences in outcomes between the two study arms, the Wilcoxon Signed-Rank test will be used. Frequencies across time will be assessed via the McNemar Test for Proportions. All statistical tests will be two-sided, with a significance level of 0.05.

Goals and milestones will be rigorously evaluated each quarter and adjustments made if/when we are behind our target. As one example, we expect to enroll 25 new participants, or 25% of our total goal, into the AI every quarter of the first year. If, for some reason, we are only able to recruit 10% of the total participants after the first quarter, we will adjust our methods of recruitment, send out an additional mailing to Housing Choice Voucher residents and pursue real-time monitoring of eligible patients in our health system to ensure that we are reaching all adults who need our program. If after those efforts we've only met 30% of our recruitment goal after the second quarter, we may propose a limited expansion in our targeted area, but we do not foresee this being an issue.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Resident of targeted Southwest or Westside communities of Chicago
* Diagnosed with asthma by a health care provider
* Has poorly controlled asthma, meeting one of the following criteria: Hospitalized for asthma within 12 months preceding enrollment; Visited an ED for asthma within 12 months preceding enrollment; Symptoms of persistent asthma - has been prescribed an inhaled corticosteroid in the last year, has asthma symptoms > 2 days/week over past 2 months, has nighttime symptoms 3-4 times/month or more, or Short acting beta2-agonist use for symptom control >2 days/week; or Has poorly controlled asthma per the Asthma Control Test (i.e., ACT score < 19)
* Has completed the HCWABT Active Intervention

Exclusion Criteria:

* Participated in another comprehensive asthma program within the past year
* Plans to move out of Chicago within the study period
* Has a diagnosis of Chronic Heart Failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of Emergency Department Visits | 12 months
  Number of visits to an emergency department in prior 12 months
Daytime asthma symptom frequency | 12 months
  Average frequency of daytime asthma symptoms over the past 12 months
Asthma-related quality of life score | 12 months
  Score on asthma-related quality of life questionnaire

SECONDARY OUTCOMES:
Asthma Control Test score | 12 months
  Score on Asthma Control Test
Activity-limited days | 12 months
  Number of self-reported activity-limited days
Access to medical care | 12 months
  Self-reported access to primary care physician, insurance coverage, and medications

CONTACTS AND LOCATIONS:
Overall Officials: Helen Margellos-Anast, MPH, Principal Investigator — Sinai Health System
Locations (1):
- Mount Sinai Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No